CLINICAL TRIAL: NCT05541341
Title: Effectiveness and Safety of Tisagenlecleucel Therapy in Brazilian Patients With B-lymphocyte Malignancies: a 15-year Prospective Registry Study on Three Cohorts.
Brief Title: Effectiveness and Safety of Tisagenlecleucel Therapy in Brazilian Patients With B-lymphocyte Malignancies
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019BBR02
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-cell Lymphoma; Acute Lymphoblastic Leukemia; Follicular Lymphoma
Keywords: Diffuse Large B-cell Lymphoma; DLBCL; Acute Lymphoblastic Leukemia; ALL; Tisagenlecleucel; Brazil; NIS; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular | interventions — tisagenlecleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (3):
- Acute Lymphoblastic Leukemia (ALL): Children/young adult patients with relapsed/refractory B-cell acute lymphoblastic leukemia who received tisagenlecleucel infusion
  Interventions: Other: tisagenlecleucel
- Diffuse Large B-cell Lymphoma (DLBCL): Adult patients with relapsed/refractory Diffuse Large B-cell Lymphoma who received tisagenlecleucel infusion
  Interventions: Other: tisagenlecleucel
- Follicular Lymphoma (FL): Patients of any gender aged 18 year or older, with relapsed/refractory Follicular Lymphoma who received tisagenlecleucel infusion.
  Interventions: Other: tisagenlecleucel

INTERVENTIONS:
Other: tisagenlecleucel — Prospective observational study. There is no treatment allocation. Patients prescribed with tisagenlecleucel in the commercial setting or out-of-specification (OOS) are eligible to enroll into this study

SUMMARY:
This will be a multicenter, national, non-interventional, prospective cohort study

DETAILED DESCRIPTION:
Eligible participants will be pediatric (<18 years) and adult patients (aged 18 years or older) with B-cell malignancies who have received tisagenlecleucel through the commercial setting or out-of-specification (OOS) use in Brazil. We will collect data prospectively and complement missing information with retrospective data collection, when necessary. It is anticipated that approximately 200 patients will be enrolled in the cohort over 5 years divided among the study indications.

Since this is a non-interventional study, no administration of study drug or application of questionnaires will be mandated by this protocol. The study will consist of a "Pre-infusion" and a "Post infusion follow-up period" for up to 15 years post tisagenlecleucel infusion. All patients will be followed until death or last scheduled visit, whichever comes first.

For the study, "pre-infusion" and "follow-up post infusion" phases are defined as:

* "Pre-infusion" will consist of the patient's information from the time of diagnosis untiljust prior to infusion with tisagenlecleucel.
* "Follow-up Post infusion" information will comprise any information from the infusionof tisagenlecleucel onwards.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet the following criteria:

1. Patients who receive tisagenlecleucel infusion in the commercial setting or out-of-specification (OOS) use, AND
2. Signed informed consent must be obtained prior to participation in study, AND

   For ALL participants:
3. Patients of any gender aged 0-17 years (named as pediatric) with relapsed/ refractory B-cell ALL diagnosis that received tisagenlecleucel infusion, OR
4. Patients of any gender, aged 18-25 years (named as adults) - with relapsed/ refractory B-cell ALL diagnosis that received tisagenlecleucel infusion, OR

   For DBLCL and FL participants:
5. Patients of any gender aged 18 years or older, who have been diagnosed with relapsed/ refractory Diffuse Large B-cell Lymphoma and received tisagenlecleucel infusion.

Exclusion Criteria:

1. Patients who did not consent to data collection.
2. Patients who received tisagenlecleucel infusion as part of any interventional clinical trial.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include pediatric/ adult patients with relapsed/refractory B-cell acute lymphoblastic leukemia aged 0-25 years and adult patients aged ≥ 18 years with relapsed/refractory Diffuse Large B-cell Lymphoma and relapsed/refractory follicular lymphoma, who received tisagenlecleucel infusion in the commercial setting or out-of-specification.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2043-11-23 (Estimated); Study Completion 2043-11-23 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 15 years
  The overall response rate will be defined as the total proportion of participants exhibiting either the best overall response (BOR) of complete or partial responses and the proportion of patient with BOR of CR/PR or CR/CRi for ALL patients will be reported along with its 95% CI.
  For ALL participants, the BOR will be defined as a CR or a CRi in accordance with National Comprehensive Cancer Network (NCCN) guidelines and previous guidelines (Appelbaum et al 2007)(Cheson et al 2003).
  For lymphomas, the BOR will be defined as a CR or PR in accordance with the Cheson response criteria (Cheson et al 2007) and the Lugano classification (Cheson et al 2016).
MRD negative overall response rate | Up to 15 years
  The percentage of B-cell ALL patients who achieve a Best Overall Response (BOR) of CR or CRi with a Minimal residual disease (MRD) negative bone marrow will be provided with 95% CI.
Duration of overall response (DOR) | Up to 15 years
  Duration of overall response (DOR) applies only to patients whose best overall disease response was either:
  * CR or PR for patients with lymphomas, or
  * CR or a CRi for patients with ALL.
  DOR will be defined as the time from the date of first documented disease response (Complete Response (CR) or PR for patients with lymphomas, and Complete Remission (CR) or CRi for patients with ALL), whichever occurs first, to the date of first documented progression or first documented relapse according to indication, or to the date of death due to the underlying disease.
  In case a patient does not have progression/relapse or death due to underlying disease (defined as the event for this outcome) prior to data cut-off, DOR will be censored at the date of the last assessment on or prior to the earliest censoring event.
Relapse-free survival (RFS) | Up to 15 years
  RFS is measured by the time from date of first documented disease response as CR or CRi to relapse or death due to any cause in ALL patients.
  In case a patient does not have relapse or death due to any cause prior to data cutoff, RFS will be censored at the date of the last adequate assessment on or prior to the earliest censoring event.
Event-free survival (EFS) for ALL patients | Up to 15 years
  EFS is the time from date of first tisagenlecleucel infusion to treatment failure, relapse or death from any cause, whichever occurred first, for B-cell ALL patients.
Progression free survival (PFS) for DLBCL patients | Up to 15 years
  PFS is defined as the time from the date of first infusion to the date of event defined as the first documented progression of lymphoma or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of the last adequate assessment.
  In case a patient does not have progression or death prior to data cutoff, PFS will be censored at the date of the last adequate assessment on or prior to the earliest censoring event.
Overall survival (OS) | Up to 15 years
  Overall survival is the time from date of first tisagenlecleucel infusion to the date of death due to any reason, In case a patient is alive at the date of last contact on or before data cutoff, OS is censored at the date of last contact.
Number of ALL patients with hematologic recovery | Up to 15 years
  Dates of hematological recovery (i.e., dates of Absolute Neutrophil Count (ANC) and platelet recovery) will be collected.
  ANC recovery is defined as an ANC of ≥ 0.5 × 109/L (500/mm^3) for 3 consecutive laboratory values obtained on different days. Date of ANC recovery is the date of the first of 3 consecutive laboratory values where the ANC is ≥ 0.5 × 109/L (CIBMTR).
  The first date of the 3 consecutive laboratory values obtained on different days where the platelet count was ≥ 20 × 109/L should be recorded. It should be ensured that no platelet transfusions were administered for 7 days immediately preceding this date (CIBMTR).

SECONDARY OUTCOMES:
The type and frequency of SAEs and AE of special interest | Up to 15 years
  The type and frequency of SAEs and AE of special interest (including secondary malignancies) will be collected
Incidence and severity of CRS and ICANS among HTLV 1 and 2 positive versus HTLV 1 and 2 negative patients | Up to 15 years
  Incidence and severity of Cytokine release syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) among Human T-cell Lymphotropic Virus (HTLV) 1 and 2 positive versus HTLV 1 and 2 negative patients.
  For CRS AE the protocol will follow the American Society of Transplant and Cellular Therapy (ASTCT) CRS Consensus Grading.
  For ICANS AE the protocol will follow ASTCT consensus as well. Which establishes the Immune effector Cell-associated Encephalopathy (ICE Score) for adults/ adolescents and Cornell Assessment of Pediatric Delirium (CAPD) for pediatric patients under 12 years
Pregnancy rates | Up to 15 years
  Pregnancy rates will be collected
Number of patients with confirmed secondary malignancies diagnosis | Up to 15 years
  Number of patients with confirmed secondary malignancies diagnosis will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Brazil (5):
  - Novartis Investigative Site, Minas Gerais, Belo Horizonte
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo

IPD SHARING:
Plan to Share IPD: No